CLINICAL TRIAL: NCT00892905
Title: Comparison Between Point of Care INR and aPTT Hemochron Jr Whole Blood Measurement With Standard Laboratory in Patients Having Elective First Time on Pump Coronary Artery Bypass Grafting (CABG)
Brief Title: Comparing Point of Care Clotting Tests in the OR Versus Standard Laboratory Clotting Tests
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Summer Syed, MD, Hamilton Health Sciences
Organization: McMaster University (Other)
Other Study IDs: 07-467
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-01

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: coagulation; INR; aPTT; point of care; laboratory; CABG; surgery
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POC INR and APTT Hemochron: Adult patients undergoing elective on pump coronary artery bypass grafting surgery who have not received anticoagulants or clopidogrel within 5 days preoperatively.

SUMMARY:
The purpose of this study is determine the agreement of point of care (POC) clotting tests (INR and aPTT) by the POC device by Hemochron Jr versus standard laboratory clotting tests (INR and aPTT) in patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
The study is a correlation between POC Hemochron Jr INR and aPTT with the standard.

ELIGIBILITY:
Inclusion Criteria:

* did not receive anticoagulants or clopidogrel within 5 days preoperatively

Exclusion Criteria:

* history of coagulopathy
* heparin resistance
* receiving heparin or warfarin
* hepatic or renal dysfunction
* pregnancy
* urgent or emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing elective on pump CABG
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Correlation between pre cardiopulmonary bypass (CPB) and post CPB POC INR and PTT with standard laboratory INR and PTT | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Summer Syed, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada